CLINICAL TRIAL: NCT02698566
Title: An Open-Label, Single-Arm Phase IIIb Study in Patients With Neovascular Age-Related Macular Degeneration or Macular Edema Secondary to Retinal Vein Occlusion to Evaluate the Usability of Lucentis® 0.5 mg Prefilled Syringe
Brief Title: A Study in Patients With Neovascular Age Related Macular Degeneration or Macular Edema Secondary To Retinal Vein Occlusion to Evaluate Usability of the Ranibizumab (Lucentis®) Prefilled Syringe (PFS)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: GX30020
Record Dates: First submitted 2016-02-29; First posted 2016-03-03 (Estimated); Results first posted 2017-07-26 (Actual); Last update posted 2017-09-21 (Actual); Status verified 2017-08

CONDITIONS: Macular Edema
MeSH Terms: conditions — Macular Edema | interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ranibizumab PFS (Experimental): Healthcare professionals (HCPs) will administer ITV injections of ranibizumab 0.5 mg delivered via PFS to enrolled patients (1 injection to each patient) on Day 1.
  Interventions: Drug: Ranibizumab

INTERVENTIONS:
Drug: Ranibizumab — Patients will receive single ITV injection of ranibizumab 0.5 mg delivered via PFS on Day 1.
  Other Names: Lucentis

SUMMARY:
This is a multicenter study designed to evaluate usability of ranibizumab PFS in patients with neovascular age related macular degeneration or macular edema secondary to retinal vein occlusion.

DETAILED DESCRIPTION:
The purpose of this study is to assess the ability of HCPs to follow the instructions for use (IFU) to prepare and administer a ranibizumab PFS ITV injection dose to patients.

ELIGIBILITY:
Inclusion Criteria:

Ocular

* Study eye deemed to be indicated for ranibizumab ITV therapy at the discretion of the retina specialist

Exclusion Criteria:

Concurrent Ocular Conditions

* Patients legally blind in one or both eyes
* History of or any current clinically relevant intraocular inflammation or ocular inflammatory reaction (any grading from trace and greater is excluded), including non-infectious uveitis or uveitis, or sterile inflammatory reaction after the past ITV injections with any agent
* Active disorder of ocular adnexa and skin in the study eye, including ocular surface infections
* History of or any current indication of excessive bleeding and recurrent hemorrhages, including any prior excessive intraocular (including subconjunctival) bleeding or hemorrhages after ITV injection or intraocular procedures
* Uncontrolled intraocular pressure greater than (>) 25 millimeters of mercury (mmHg) in the study eye (uncontrolled means that it occurs even with intraocular pressure-lowering therapy)
* Use of therapies that are known to be toxic to any ocular tissues within the 6 months prior to enrollment

Prior Ocular Therapies

* Treatment with any ITV injection within the 27 days prior to Day 1
* Any invasive intraocular surgery, prior long-acting therapeutic agent, or ocular drug release device implantation (approved or investigational) in the study eye at any time during the past 3 months

General

* Receipt of any systemic (non-ocular) investigational drug within 3 months prior to Day 1
* Current systemic coagulation or bleeding disorders and history of recurrent hemorrhages
* Intolerance or known reaction to prior biological therapies
* History of other diseases or physical or laboratory examination findings that per the retina specialist represent a contraindication to ranibizumab use in the patient or may represent an unwarranted patient risk.
* Uncontrolled hypertension (systolic >160 mmHg and/or diastolic >100 mmHg while sitting)
* Current systemic infectious disease or a therapy for active infectious disease
* Pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2016-03-21 (Actual); Primary Completion 2016-04-05 (Actual); Study Completion 2016-04-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (4):
- United States (4):
  - Paducah Retinal Center, Paducah, Kentucky
  - Char Eye Ear &Throat Assoc, Charlotte, North Carolina
  - Southeastern Retina Associates, Chattanooga, Tennessee
  - Charles Retina Institution, Germantown, Tennessee

REFERENCES:
- [Derived] Antoszyk AN, Baker C, Calzada J, Cummings H, So J, Quezada-Ruiz C, Haskova Z. Usability of the Ranibizumab 0.5 mg Prefilled Syringe: Human Factors Studies to Evaluate Critical Task Completion by Healthcare Professionals. PDA J Pharm Sci Technol. 2018 Jul-Aug;72(4):411-419. doi: 10.5731/pdajpst.2017.008342. Epub 2018 May 31. PMID 29853609

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participant Flow module includes the number of patients enrolled ("35") as well as the number of healthcare professionals ("3") who administered intravitreal (ITV) injections to enrolled patients.
Groups:
- Ranibizumab PFS - Patients: Healthcare professionals (HCPs) administered ITV injections of ranibizumab 0.5 milligrams (mg) delivered via PFS to enrolled patients (1 injection to each patient) on Day 1.
- Ranibizumab PFS - HCPs: HCPs administered ITV injections of ranibizumab 0.5 mg delivered via PFS to enrolled patients (1 injection to each patient) on Day 1.
Period: Overall Study
Arm/Group | Ranibizumab PFS - Patients | Ranibizumab PFS - HCPs
Started | 35 | 3
Completed | 35 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled patients.
Groups:
- Ranibizumab PFS: HCPs administered ITV injections of ranibizumab 0.5 mg delivered via PFS to enrolled patients (1 injection to each patient) on Day 1.
Arm/Group | Ranibizumab PFS
Number analyzed (Participants) | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 78.3 (6.8)
Sex/Gender, Customized [Number; unit: patients] — Gender information was not collected for this study.
  patients
    Female | 0
    Male | 0
    Unknown | 35

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Successful Task Completions
Description: Product use tasks included sequence of steps starting from opening the carton, removing contents from carton to disposing of used PFS and needle. Tasks were considered to be successfully completed if the correct results were achieved without a use error, even if the instructions for use (IFU) were not followed exactly (example: not removing the needle cap prior to adjusting a dose). Usage error was defined as user action or lack of user action while using the medical device that led to a different result than intended by the manufacturer or expected by the user. The ability of HCPs to follow the IFU to prepare and administer a ranibizumab PFS ITV injection dose to patients was evaluated by successful task completion.
Time Frame: Day 1
Population: Three HCPs referred to as 'participants' performed tasks on 35 enrolled patients by giving single PFS ITV injection to each patient. The percentages are calculated out of the total 35 PFS ITV injections administered.
Measure: Number; unit: percentage of tasks
Units Other Than Participants: ITV injections
Arm/Group | Ranibizumab PFS
Number analyzed (Participants) | 3
Number analyzed (ITV injections) | 35
percentage of tasks
  Open the carton | 100
  Remove contents from carton | 100
  Peel the lid off the blister pack | 100
  Carefully remove the PFS using aseptic technique | 100
  Snap off PFS cap | 100
  Firmly screw needle onto the Luer lock of PFS | 100
  Remove needle cap | 100
  Dose preparation: aligning stopper with dose line | 100
  Insert PFS at injection site | 100
  Slowly inject full dose | 100
  Remove PFS from injection site | 100
  Dispose of used PFS and needle | 100

2. Primary Outcome: Percentage of PFS Usage Errors on Safety Critical Tasks
Description: Usage error was defined as user action or lack of user action while using the medical device that led to a different result than intended by the manufacturer or expected by the user. Safety critical tasks where those in which use error could have a reasonably foreseeable potential for clinical impact or harm.
Time Frame: Day 1
Population: Three HCP's referred to as 'participants' performed tasks on 35 enrolled patients by giving single PFS ITV injection to each patient. The percentages are calculated out of the total 35 PFS ITV injections administered.
Measure: Number; unit: percentage of usage errors
Units Other Than Participants: ITV injections
Arm/Group | Ranibizumab PFS
Number analyzed (Participants) | 3
Number analyzed (ITV injections) | 35
percentage of usage errors | 0

3. Primary Outcome: Percentage of PFS Usage Errors on Essential Tasks
Description: Usage error was defined as user action or lack of user action while using the medical device that led to a different result than intended by the manufacturer or expected by the user. Essential tasks were those that were required in order to complete the use process for effective use of the product.
Time Frame: Day 1
Population: as for outcome 2
Measure: Number; unit: percentage of usage errors
Units Other Than Participants: ITV injections
Arm/Group | Ranibizumab PFS
Number analyzed (Participants) | 3
Number analyzed (ITV injections) | 35
percentage of usage errors | 0

ADVERSE EVENTS:
Time Frame: Day 1 to Day 7
Description: No safety analyses were pre-specified as objectives in study GX30020. However, in accordance with Good Clinical Practices (GCP) guidelines, adverse events and serious adverse events that occurred during the 7-day study-reporting period were monitored and reported in this section.
Arm/Group | Ranibizumab PFS
Serious Adverse Events (participants affected / at risk) | 0/35
Other Adverse Events (participants affected / at risk) | 1/35
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ranibizumab PFS (N=35)
Conjunctival hemorrhage (Eye disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.